CLINICAL TRIAL: NCT06276790
Title: The Predictive Value of an Ultrasound Quantitative Scoring System for Treatment Method Selection in Patients With Caesarean Scar Pregnancy: A Single-Centre Retrospective Study
Brief Title: Objective Analysis of Caesarean Scar Pregnancy
Status: Completed | Type: Observational
Sponsor: Chengde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Jianwen Du, physician, Chengde Central Hospital
Other Study IDs: ChengdeCentralHospital
Record Dates: First submitted 2024-01-25; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Caesarean Scar Pregnancy; Ultrasound Scoring System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-risk group
  Interventions: Procedure: ultrasound-guided/hysteroscopic curettage
- high-risk group
  Interventions: Procedure: Procedure/Surgery: laparoscopic removal of the pregnancy lesion

INTERVENTIONS:
Procedure: ultrasound-guided/hysteroscopic curettage — ultrasound-guided/hysteroscopic curettage
  Groups: low-risk group
Procedure: Procedure/Surgery: laparoscopic removal of the pregnancy lesion — laparoscopic removal of the pregnancy lesion
  Groups: high-risk group

SUMMARY:
This study uses a systematic scoring method combined with clinical and ultrasound data to comprehensively evaluate patient conditions and explore the guiding value of the ultrasound quantitative scoring system for selecting the surgical approach for caesarean scar pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* history of at least one previous caesarean section
* symptoms suggestive of caesarean scar pregnancy, such as unexplained abnormal vaginal bleeding, abdominal pain, cervical pain or abnormal uterine activity during pregnancy
* amenorrhea ≤84 days
* ultrasound examination suggesting a single gestational sac with intact morphology
* stable maternal vital signs

Exclusion Criteria:

* mass-type caesarean scar pregnancy
* previous medication or surgical treatment before ultrasound examination
* haemodynamically unstable patients
* patients with surgical contraindications
* incomplete or lost follow-up clinical data
* patients with severe medical conditions such as hypertension, diabetes, hyperthyroidism and haemophilia

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: A total of 117 patients with caesarean scar pregnancy admitted to the Obstetrics and Gynecology Inpatient Area of Chengde Central Hospital, China, from January 2019 to December 2022 were selected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during surgery
  The patient's blood loss during surgery. Check the blood volume in ml of the aspirator reservoir.
length of hospital stay | Within 1 week
  Number of days the patient was hospitalized. Discharge assessment: vital signs stable, no abdominal pain, no active bleeding.
serum β-HCG levels | Within 2 weeks after the operation
  The time taken for serum β-HCG levels to return to normal

CONTACTS AND LOCATIONS:
Locations (1):
- Chengde Central Hospital, Chengde, China